CLINICAL TRIAL: NCT00829062
Title: Presenting Evidence Based Practice to an Insurance Provider to Expand Coverage of Continuous Subcutaneous Insulin Infusion (CSII) in Pediatric Patients With Diabetes
Brief Title: Expanding Coverage of Continuous Subcutaneous Insulin Infusion in Pediatric Patients With Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants met inclusion criteria.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Amanda G. Fridlington, CPNP, Pediatric Nurse Practitioner- Children's Mercy Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 08-11-178E
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Insulin pump; Glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucose sensor (No Intervention): Children who have assented to wear a 72 hour physician ordered continuous glucose monitor.
  Interventions: Device: Continuous glucose glucose sensor- physician ordered

INTERVENTIONS:
Device: Continuous glucose glucose sensor- physician ordered — Charts will be reviewed to identify recipients of Missouri Medicaid who receive daily injections to manage their diabetes. Children who have submitted an application for the Medtronic MiniMed insulin pump will be identified by the PI and Medtronic Diabetes. They will be asked to wear a 72 hour continuous glucose monitor. The children who wear the sensor will be asked to keep a daily logbook of their blood sugars, activities, food intake, and insulin doses during this 72 hour period. The families of the children will be provided with a pre-addressed FedEx envelope for them to return the digital recorder and daily logbooks to the PI. The results of the glucose sensor will be downloaded by the PI. The families will be contacted by the PI with the results and treatment recommendations.
  Other Names: Glucose sensor; Continuous glucose sensor; Physician ordered glucose sensor

SUMMARY:
The purpose of the study is to present evidence based literature and clinical data to the medical directors at Missouri Medicaid to help modify the existing policy regarding insulin pump therapy in pediatric patients with diabetes.

DETAILED DESCRIPTION:
Results from the Diabetes Control and Complications Trial (DCCT) showed that more aggressive and intensive management of diabetes leads to a reduction in the incidence of diabetes related complications in adolescents and adults. Therefore, early initiation of intensive insulin regimens that have been proven to normalize blood sugars as much as possible need to be initiated in youth with type 1 diabetes mellitus (T1DM) to improve outcomes in adulthood. However, despite this understanding, there remains no consensus for how to best manage insulin delivery in children diagnosed with T1DM.

Intensive insulin treatment of diabetes typically entails one of two therapies: MDI (multiple daily injections) or CSII also know as insulin pump therapy. MDI requires several insulin injections per day to achieve near normal glycemic control which can also lead to a subsequent increased risk of severe hypoglycemia. The insulin pump allows the user to program in various basal insulin rates, as low as 0.025 units/hr, throughout the day and night to better match one's physiologic insulin secretion, and eliminates the need for insulin injections throughout the day.

Management of T1DM in the pediatric setting presents several challenges for the patient, caregivers, and health care providers. Children and adolescents tend to have wide fluctuations in their blood glucose levels due to varying amounts of physical activity from day to day. Additionally, infants, toddlers, and school age children have eating habits that are very unpredictable and often eat small quantities making it quite difficult to accurately administer small doses of insulin through an insulin syringe or pen device. Finally, there is increasing evidence to support that infants and toddlers who experience severe hypoglycemia may have resultant neurologic deficits. Previous research has demonstrated that pediatric patients on insulin pump therapy had better glycemic control when compared to pediatric patients who were managed on MDI alone. Patients on insulin pumps and their parents have reported more flexibility with meals and daily activities, lower hemoglobin A1c levels, decreased variability in blood sugar readings, and fewer episodes of hypoglycemia.

Despite the vast research documenting the benefits of insulin pump therapy, some insurance companies continue to be hesitant in covering CSII in pediatric patients with diabetes. The findings from this study and supporting evidence will be presented to medical directors at Missouri Medicaid to help expand coverage of CSII in pediatric patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 months-17 years old diagnosed with Type I Diabetes Mellitus receiving diabetes care at Children's Mercy Hospital
* Patients/families must be able to read and speak English
* Patients will need to have had a minimum of 3 clinic visits over the past year
* Patients who are recipients of Missouri Medicaid that have been denied or are awaiting Medtronic MiniMed insulin pump coverage
* Patients receiving insulin injections

Exclusion Criteria:

* Non Missouri Medicaid patients on insulin injections
* Recipients of Missouri Medicaid who are currently on insulin pump therapy

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
The aim of this project is to present evidence based practice to Missouri Medicaid to expand coverage of continuous subcutaneous insulin infusion (CSII) in pediatric patients with diabetes. - Hemoglobin A1C | 12 months

SECONDARY OUTCOMES:
Glycemic variability as shown by continuous glucose recording | 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Amanda G Fridlington, MSN, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Boland EA, Grey M, Oesterle A, Fredrickson L, Tamborlane WV. Continuous subcutaneous insulin infusion. A new way to lower risk of severe hypoglycemia, improve metabolic control, and enhance coping in adolescents with type 1 diabetes. Diabetes Care. 1999 Nov;22(11):1779-84. doi: 10.2337/diacare.22.11.1779. PMID 10546007
- [Background] Ramchandani N, Ten S, Anhalt H, Sinha S, Ching J, Finkelstein A, Maclaren NK. Insulin pump therapy from the time of diagnosis of type 1 diabetes. Diabetes Technol Ther. 2006 Dec;8(6):663-70. doi: 10.1089/dia.2006.8.663. PMID 17109598
- [Background] Shalitin S, Phillip M. The role of new technologies in treating children and adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2007 Oct;8 Suppl 6:72-9. doi: 10.1111/j.1399-5448.2007.00279.x. PMID 17727388
- [Background] Weinzimer SA, Ahern JH, Doyle EA, Vincent MR, Dziura J, Steffen AT, Tamborlane WV. Persistence of benefits of continuous subcutaneous insulin infusion in very young children with type 1 diabetes: a follow-up report. Pediatrics. 2004 Dec;114(6):1601-5. doi: 10.1542/peds.2004-0092. PMID 15574621